CLINICAL TRIAL: NCT01352897
Title: A Registry to Collect Data of Efficacy and Safety Between Rosuvastatin, and Atorvastatin and Simvastatin In Subjects With Type IIa and IIb Hypercholesterolaemia Under Real Clinical Settings
Brief Title: Registry On Efficacy and Safety Of Rosuvastatin, and Atorvastatin and Simvastatin In Hypercholesterolaemia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca Singapore
Other Study IDs: NIS-CSG-CRE-2011/1
Record Dates: First submitted 2011-05-09; First posted 2011-05-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Hypercholesterolaemia
Keywords: Cholesterol; rosuvastatin; retrospective
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this follow-up retrospective study is to evaluate the long term efficacy and safety of rosuvastatin in reducing lipid parameters in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Primary hypercholesterolemia
* Subjects from first rosuvastatin Registry study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from primary care and specialist clinics
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who maintain US NCEP ATP III LDL-C target goals after long-term therapy | Up to 8 years

SECONDARY OUTCOMES:
LDL-cholesterol levels | Up to 8 years
HDL-cholesterol levels | Up to 8 years
Proportion of patients having raised levels of serum CK or ALT | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: DR ARTHUR TAN, MBBS, Principal Investigator — ARTHUR TAN HEART CLINIC, GLENEAGLES MEDICAL CENTRE
Locations (1):
- Research Site, Singapore, Singapore